CLINICAL TRIAL: NCT03617146
Title: Coaching and Education for Diabetes Distress: a Randomized Controlled Trial (CEDD Trial)
Brief Title: Coaching and Education for Diabetes Distress
Acronym: CEDD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Charles C Chima, Adjunct Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 52960-I
Record Dates: First submitted 2018-07-27; First posted 2018-08-06 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Distress
Keywords: Diabetes Distress; Diabetes Mellitus; Diabetes Control; Health Coaching; Diabetes Self-management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Two-arm parallel randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the behavioral intervention, neither participants nor clinic staff can be blinded to allocation. However, to avoid bias in assessing outcomes, the analyst who will abstract the outcomes data from the electronic health record will not have access to information about the allocation. Hence retrieval of data on baseline and follow up diabetes distress scores, HbA1c, and diabetes self-management behaviors, and the creation of the analysis dataset will be done without knowledge or consideration of allocation status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants in the intervention arm will receive the following interventions:
  Month 1: Diabetes Distress-specific Education.
  Months 1 to 3: Six 30 to 45-minute telephone-based health coaching sessions targeting diabetes distress reduction and self-care improvement.
  Month 3: Follow up distress-specific education.
  Months 4 and 5: Two 30 to 45 minute telephone-based health coaching sessions targeting diabetes distress reduction and self-care improvement.
  Interventions: Behavioral: Health coaching; Other: Diabetes Distress-specific Education
- Control Arm (Active Comparator): Participants in the control arm will receive the following interventions:
  Month 1: Diabetes Distress-specific Education (same as for the intervention arm).
  Month 3: Follow up distress-specific education (same as for the intervention arm).
  Interventions: Other: Diabetes Distress-specific Education

INTERVENTIONS:
Behavioral: Health coaching — The intervention will seek to help participants express their diabetes emotional needs and to work with them to figure out what can be done to meet those needs. Depending on the unique needs of each participant, the coaching approach for this study will include: improving motivation and self-efficacy for diabetes management using motivational interviewing and appreciative inquiry; building trust and rapport through mindful listening, open-ended inquiry, and perceptive reflections; and expressing empathy through nonviolent communication. Each participant will receive eight individual coaching sessions over a five month period. All coaching sessions will be delivered over the phone (i.e. telecoaching). The coaching intervention will be done by a certified health and wellness coach.
  Other Names: Telecoaching
  Arms: Intervention Arm
Other: Diabetes Distress-specific Education — A diabetes distress-specific education that explains what diabetes distress is, why it matters, and its four domains. In addition, the participant is given feedback on his or her distress score and advised on ways to deal with the areas of greatest distress. Participant is linked with resources to overcome any expressed needs. The education is provided by a trained medical assistant.

SUMMARY:
Diabetes distress (DD) is a negative emotional reaction to a diagnosis of diabetes and concerns about the burden of managing diabetes, the risk of complications, and inadequate support system. DD is common among people with diabetes and is strongly associated with poor diabetes self-care and poor diabetes control. Reducing DD should thus be an important component of diabetes management. In line with the growing evidence, the American Diabetes Association now recommends that providers "routinely monitor people with diabetes for diabetes distress, particularly when treatment targets are not met". Despite increased recognition of the need to manage DD, interventions that are both feasible and effective for reducing DD in routine care settings are not yet known. A pilot study showed that health coaching (HC) has some efficacy in addressing DD but no adequately powered study has implemented a pragmatic research design capable of assessing the real-world effectiveness of HC in reducing DD.

This study seeks to assess whether HC effectively reduces DD among primary care patients with diabetes, and whether HC is more effective than an educational program targeting DD. The investigators hypothesize that over a 6-month period, patients with poorly controlled diabetes and DD who enroll in and complete at least five HC sessions will achieve higher and clinically significant reductions in DD and HbA1c, and greater compliance with diabetes self-care recommendations than those who receive only an educational program targeting DD as part of usual diabetes care.

The two-arm randomized controlled trial for patients with poorly-controlled diabetes is taking place at an academic family medicine practice in Houston, Texas. Both arms will receive usual care, which includes education about DD. In addition, the intervention arm will receive eight HC sessions over a five-month period. The primary outcome measure is reduction in DD over a six month period. Additional outcome measures include changes in glycemic control (HbA1C) and self-care practices (medication adherence, dietary, and physical activity behaviors). The study will also measure satisfaction and willingness-to-pay for HC to determine the extent to which HC, if effective for reducing DD, can be operationalized in similar healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Has had a diagnosis of type 2 diabetes for at least 6 months
* Aged 18 to 75 years
* Most recent HbA1c taken within 30 days was ≥ 8.0
* At least moderate diabetes distress (a mean score ≥ 2.0 on the 17-item Diabetes Distress Scale).

Exclusion Criteria:

* Moderately-severe to severe depression: Patient Health Questionnaire (PHQ9) score ≥15
* Other severe mental health disorder (e.g. Alzheimer's, schizophrenia)
* Current pregnancy
* Severe diabetes complications or functional deficits (e.g. kidney failure requiring dialysis, amputation, blindness).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Diabetes distress score | 3 months and 6 months from baseline
  Change in diabetes distress score as measured by the diabetes distress scale (DDS). DDS scores range from 1 to 6, with scores that are less than 2.0 being indicative of little or no distress. Hence scores of 2.0 and above are significant and higher values are indicative of worse outcome.

SECONDARY OUTCOMES:
HbA1c | 3 months and 6 months from baseline
  Change in glycemic control as measured by HbA1c
Self-care behaviors (medication adherence, dietary practices, and physical activity behaviors) | 3 months and 6 months from baseline
  Change in medication adherence, dietary practices, and physical activity behaviors, as measured by the respective medication, diet, and exercise subscales of the Summary of Diabetes Self-Care Activities (SDSCA) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Chima, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor Family Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Chima CC, Salemi JL, Sidani MA, Zoorob RJ. Coaching and Education for Diabetes Distress (CEDD): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Apr 2;8(4):e12166. doi: 10.2196/12166. PMID 30938687